CLINICAL TRIAL: NCT05467371
Title: Safe Babies Parenting Action Plan RCT
Brief Title: Safe Babies: Parenting Action Plan ( PAP )
Acronym: PAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Dorothy Mandell, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-SPH-23-1042
Record Dates: First submitted 2022-07-15; First posted 2022-07-20 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Parenting; Motivational Interviewing; Maltreatment/Abuse
Keywords: parenting education; maternal mental health; infant maltreatment; motivational interviewing

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled trial with maternal caregivers of infants 2 months and younger. Maternal caregivers who consent to be in the study will be randomized into one of two groups. One group will get Safe Kids home safety education and the other group will receive the Parenting Action Plan with motivational interviewing techniques.
Who Masked: Outcomes Assessor
Masking Description: All data will be blinded prior to analysis. The outcomes assessor will not know study allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Parenting Action Plan (Experimental): The parenting action plan is a booklet with information that focuses on sleep hygiene, soothing a crying baby, what to do when the baby's crying is overwhelming, identifying safe caregivers in case of emergency, and issues surrounding feeding and bonding with the baby. Maternal caregivers will receive the booklet via mail and a trained research staff member will virtually go over the booklet using motivational interviewing strategies
  Interventions: Behavioral: Parenting Action Plan
- Safe Kids Home Safety Checklist (Active Comparator): The Safe Kids Home Safety Checklist is a handout with information that focuses on home safety for parents of young children. Maternal caregivers will receive the handout via mail and a trained research staff member will virtually go over the handout with the parent using educational strategies.
  Interventions: Behavioral: Safe Kids Home Safety Checklist

INTERVENTIONS:
Behavioral: Parenting Action Plan — The parenting action plan a booklet with information that focuses on sleep hygiene, soothing a crying baby, what to do when the baby's crying is overwhelming, identifying safe caregivers in case of emergency, and issues surrounding feeding and bonding with the baby.
  Arms: Parenting Action Plan
Behavioral: Safe Kids Home Safety Checklist — Safe Kids created a home safety checklist to help keep kids safe, room by room.
  Arms: Safe Kids Home Safety Checklist

SUMMARY:
The goal is to examine the efficacy of the Parenting Action Plan (PAP), a booklet with information that focuses on sleep hygiene, soothing a crying baby, what to do when the baby's crying is overwhelming, identifying safe caregivers in case of emergency, and issues surrounding feeding and bonding with the baby.

DETAILED DESCRIPTION:
The purpose of this project is to evaluate whether prevention education using motivational interviewing focused on promoting positive maternal mental health, coping with inconsolable crying, life stress reduction, and positive coping strategies with difficult infant behavior can provide complimentary messaging that supports positive parental behavior and reduces risks associated with poor mental health and infant maltreatment. The goal is to examine the efficacy of the Parenting Action Plan (PAP), a booklet with information that focuses on sleep hygiene, soothing a crying baby, what to do when the baby's crying is overwhelming, identifying safe caregivers in case of emergency, and issues surrounding feeding and bonding with the baby. It is delivered using motivational interviewing techniques. This study is not designed to develop education for "at-risk" individuals, rather the purpose is to develop a populationlevel prevention program.

ELIGIBILITY:
Inclusion Criteria:

* maternal caregivers of infant 2 months and younger
* can read and speak English or Spanish
* has zoom / teams / facetime / google hangout capability

Exclusion Criteria:

* infant is older than 2 months of age
* under 18 years of age
* no video/virtual capability

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 283 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Parental Attributions change from 6 to 12 weeks post intervention | 6 and 12 weeks post intervention
  The Parent Attribution Test will be used to assess maltreatment risk. This survey was chosen because it has been shown to be predictive of maltreatment in high risk families27. Further, this survey is relatively immune to social desirability bias28, partially because it does not specifically ask parents about their own parenting practices.
Parental competency change from 6 to 12 weeks post intervention | 6 and 12 weeks post intervention
  Parental competency will be measured using the Infant Characteristics Questionnaire29. The Infant Characteristics Questionnaire measures infant temperament. It is being included because difficult infants can impact how parents assess their own parental competency. Further, "difficult" infants are also at a higher risk for maltreatment. This measure will allow us to assess whether the PAP can help increase self-assessed competency, but also whether these self-assessed competencies increase for mothers who have infants that are more "difficult."
Maternal depression change from 6 to 12 weeks post intervention | 6 and 12 weeks post intervention
  All women will be screened for depression using the Edinburg Postnatal Depression Scale34. It is important to clarify that the mothers will be screened for the study separate from the screening she will receive in the clinic. We will be assessing depression risk separately so that the medical record will not need to be used for research, nor will research information be used to inform medical decisions.
Maternal bonding change from 6 to 12 weeks post intervention | 6 and 12 weeks post intervention
  This self-report measure assesses how the parent feels about their infant and is a proxy for bonding.
Cognitive stimulation in the home change from 6 to 12 weeks post intervention | 6 and 12 weeks post intervention
  StimQ-I is a 43 point scale for measuring cognitive stimulation in the homes of infants ages 5 to 12 months. It is based on a questionnaire that is administered to the child's primary caregiver.

SECONDARY OUTCOMES:
Assess patient's Satisfaction level with the educational resource | Immediately post intervention
  Questionnaire developed to assess the parent's satisfaction with the resource

CONTACTS AND LOCATIONS:
Overall Officials: Dorothy Mandell, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (3):
- United States (3):
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Texas Health Science Center at Tyler, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No